CLINICAL TRIAL: NCT06200376
Title: A Clinical Study of Safety and Efficacy of T3011 Administered Via Intraperitoneal Injection as a Single Agent in Patients With Malignant Ascites Induced by Advanced Colorectal Cancer
Brief Title: A Clinical Study of Intraperitoneal T3011 Given as a Single Agent in Patients With Malignant Ascites Induced by Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Meng Qiu, Prof., West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MVR-T3011-ES-EC61-MA
Record Dates: First submitted 2023-10-12; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Malignant Ascites

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T3011 (Experimental)
  Interventions: Drug: T3011

INTERVENTIONS:
Drug: T3011 — T3011 will be administered intraperitoneally twice a week.

SUMMARY:
This is a prospective, open, single-arm, investigator-initiated clinical study to evaluate the safety and efficacy of intraperitoneal administration of T3011 at different doses in the treatment of malignant ascites induced by advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age ≥ 18 years and ≤ 75 years at the time of informed consent.
2. Histologically or cytologically confirmed advanced unresectable or metastatic colorectal cancer;
3. Anticipated life expectancy ≥3 months
4. Associated with medium amount of malignant ascites (defined as the amount of ascites ≥3cm by B ultrasonography in lying position accompanied by clinical symptomes like abdonimal distension and cytology tests possitive for tumor in ascites); No paracentesis performed with 28 days before first dosing; and the ascites can not be controlled by SOC according to PI judgement.
5. ECOG performance status 0-2 (including threshold);
6. Weight ≥40kg
7. Hematology:

   * White blood cell (WBC) ≥ 3.0×10^9/L;
   * Neutrophil (ANC) ≥ 1.5×10^9/L;
   * Platelet (PLT) ≥ 75×10^9/L;
   * Hemoglobin (Hb) ≥ 8.0g/dL
8. Hepatic and renal function:

   * Total bilirubin ≤ 1.5 × ULN;
   * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 × ULN for patient without liver metastasis, ≤ 5 × ULN for patients with liver metastasis;
   * Serum creatinine ≤ 1.5×ULN, or creatinine clearance ≥ 50 mL/min as determined by the Cockcroft-Gault equation;
   * Abumin≥30 g/L
9. Coagulation:

   * INR≤1.5 x ULN;
   * APTT≤1.5 x ULN;
10. For women of childbearing potential (WCBP), serum pregnancy test should be negative within 14 days before dosing. WCBP patients, as well as male patients with partners of WCBP, should consent to use at least one medically approved contraceptive method (e.g. surgical sterilization, oral contraceptives, intrauterine devices, abstinence or barrier contraception combined with spermicides) during the study and for at least 6 months after the last dosing;
11. Willingness to attend this study, to sign informed consent, to have good compliance, and to cooperate with follow-up visit.

Exclusion Criteria:

1. Previously diagnosed with decompensated cirrhosis, and with portal vein and branch involvement or cancer embolus;
2. Pregnant or lactating, or plan to pregnant or give birth during the trial;
3. Persistent or active infection that are not controlled by treatment including but not limited to: active tuberculosis, non-negative HIV antibody, HBsAg positive and HBV DNA ≥LOQ, HCV ab positive and HCV DNA ≥LOQ;
4. Patients with imageological confirmed brain metastasis or brain metastasis history (except patients with stable disease within 3 months before screening and not require systemic glucorticoid therapy according to PI), pia meningeal disease, spinal cord compression;
5. Autoimmune disease or related symptoms, or previously suffered from autoimmune disease;
6. History of splenectomy or organ transplantation;
7. Prior treatment with Oncolytic virus (OV) (including but not be limited to T-VEC, T3011), gene therapy, cellular therapy or tumor vaccines;
8. Requires oral or intravenous therapy against herpes virus (including but not limited to acyclovir, valaciclovir, penciclovir, famciclovir, ganciclovir, foscarnet, cidofovir). Topical use of drugs (eg. external use) are allowed;
9. Patients are scheduled to receive other therapy against malignant ascites (including but not limited to chemotherapy, target therapy, immunotherapy), and the best supportive treatment for malignant ascites is permitted (e.g., albumin supplements, etc.);
10. Patients with a known psychiatric disorder that would interfere with cooperation with the requirements of the trial;
11. History of narcotics (recreational use) and substance abuse (including alcohol) within 1 year prior to signing informed consent;
12. History of allergic reactions attributed to compounds of similar biological composition to HSV-1, IL-12, or anti-PD-1 monoclonal antibody or any excipients for T3011;
13. History or evidence of high risk cardiovascular disease, including but not limited to:

    * Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, II-III degree atrioventricular block, QT interval corrected using the Fridericia formula (QTcF) ≥ 450 msec (male) or ≥ 470 msec (female);
    * Acute myocardial infarction, unstable angina pectoris, or stroke occurred within 6 months before the first administration of the experimental drug;
    * Coronary angioplasty or stent implantation within 6 months prior to first administration of the experimental drug;
    * Rating of heart function as defined by the New York Heart Association (NYHA) standards>grade II; Cardiac valve abnormalities recorded by echocardiography (≥ grade 2). Note: Subjects with grade 1 cardiac valve abnormalities (such as mild regurgitation/stenosis) were admitted, but subjects with moderate valve thickening were excluded;
    * Left ventricular ejection fraction (LVEF) < the center lower limit. If no lower limit existed, LVEF<50%;
    * Poor blood pressure control after antihypertensive treatment (i.e. systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg);
14. History of another malignant tumor, except the following:

    * Undergo potentially curative therapy and for ≥5 years prior to the first dose of study treatment and no malignancies with known active disease and low potential recurrence risk;
    * Adequately treated non-melanoma skin cancer or lentigo with no evidence of malignancy;
    * Adequately treated carcinoma in situ without evidence of disease;
15. Received live and attenuated vaccines within 4 weeks prior to initiation of study treatment, or plan to be vaccined during the study;
16. Previous history of immunotherapy induced non-infectious pneumonitis/ interstitial lung disease (including but not limited to ≥3 grade irAE) or intolerance to immunotherapy (including but not limited to anti-PD-(L)1 monoclonal Ab), except endocrine-related irAE that can be stably controlled by hormone replacement therapy;
17. Unexplained >38.5℃ fever (except for tumor induced fever judged by PI) occurs during the screening period, baseline period or on the day of administration, which in the judgment of investigator, would interfere with patient participation in the study or patient's efficacy evaluation;
18. Any condition that PI considered may confuse the trial results, interfere with the participant's participation in the trial, or is not in the participant's best interest to participate in the trial, or a history of treatment or laboratory abnormalities, or other ineligibility for enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Adverse event | 28 days after EOT
  To evaluate the safety of intraperitoneal T3011 in the treatment of patients with malignant intraperitoneal ascites

SECONDARY OUTCOMES:
Overall response rate (ORR) | From 4th dosing to disease progression, consent withdraw, death or end of study, assessed up to 24 months
  To evaluate the ORR of intraperitoneal T3011 in the treatment of patients with malignant intraperitoneal ascites using B ultrasonography and CT scan
Disease control rate (DCR) | From 4th dosing to disease progression, consent withdraw, death or end of study, assessed up to 24 months
  To evaluate the DCR of intraperitoneal T3011 in the treatment of patients with malignant intraperitoneal ascites using B ultrasonography and CT scan
Time to onset of therapeutic paracentesis | From 4th dosing to disease progression, consent withdraw, death or end of study, assessed up to 24 months
  To evaluate the effect of intraperitoneal T3011 on the interval of therapeutic abdominal paracentesis in patients with malignant ascites
Overall survival (OS) | Up to 24 months
  To evaluate the OS of intraperitoneal T3011 in the treatment of patients with malignant intraperitoneal ascites
Quality of life questionnaire (QLQ-C30) | Up to 24 months
  The EORTC Core Questionnaire (QLQ-C30) is widely used to measure quality of life in oncology. For self-reported general health and psychological distress, a higher score indicated worse health.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China